CLINICAL TRIAL: NCT00682279
Title: A Phase I, Open-label Study of the Safety, Tolerability, and Pharmacokinetics of Oral Topotecan in Combination With Lapatinib in Subjects With Advanced Solid Tumors
Brief Title: A Phase I Study Of Oral Topotecan And Lapatinib In Subjects With Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Cancelled before enrollment
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPT109098
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Advanced Solid Tumors
Keywords: lapatinib; GW572016; topotecan; oral topotecan; SK&F-104864; EGFR; ErbB1; HER-2/neu; ErbB2; BCRP
MeSH Terms: interventions — Topotecan; Lapatinib

ARMS (1):
- This is a single-arm, dose escalation (No Intervention): This is a single-arm, dose escalation, Phase I study in which doses of oral topotecan will be escalated and lapatinib will be given initially as a fixed dose. This study will examine oral topotecan administered on a five-consecutive day schedule in combination with daily lapatinib. This study will be conducted in two parts. Part 1 of the study will investigate the impact of lapatinib on the bioavailability of oral topotecan (bioavailability phase) and Part 2 of the study will consist of dose finding to determine the MTD regimen of the combination (dose escalation phase).
  Interventions: Drug: oral topotecan (SK&F-104864); lapatinib (GW572016)

INTERVENTIONS:
Drug: oral topotecan (SK&F-104864); lapatinib (GW572016) — This is a single-arm, dose escalation, Phase I study in which doses of oral topotecan will be escalated and lapatinib will be given initially as a fixed dose. This study will examine oral topotecan administered on a five-consecutive day schedule in combination with daily lapatinib. This study will be conducted in two parts. Part 1 of the study will investigate the impact of lapatinib on the bioavailability of oral topotecan (bioavailability phase) and Part 2 of the study will consist of dose finding to determine the MTD regimen of the combination (dose escalation phase).

SUMMARY:
This is an open-label, Phase I study of oral topotecan administered in combination with lapatinib in subjects with advanced solid tumors. This Phase I study will evaluate the safety, tolerability, and pharmacokinetics of oral topotecan administered in combination with lapatinib. This study will be conducted in two parts. Part 1 of the study will investigate the impact of lapatinib on the bioavailability of oral topotecan (bioavailability phase) and Part 2 of the study will consist of dose finding to determine the maximum-tolerated dose (MTD) regimen of the combination (dose escalation phase). In Part 2 of the study, the dose of oral topotecan will be escalated while lapatinib will be given initially as fixed doses. The primary objective of the study is to determine the MTD regimen of oral topotecan administered for five-consecutive days every 21 days in combination with daily lapatinib in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide signed, written informed consent.
* Subjects must be ≥18 years of age.
* Subjects must have Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
* Subjects must have histologically or cytologically confirmed diagnosis of cancer.
* Subjects must have advanced solid malignancies without an established standard of care therapy option OR progression following the most recent therapy.
* Subjects may have measurable lesion(s) according to RECIST criteria.
* Subjects with stable CNS metastases or leptomeningeal involvement are eligible only if they are not taking oral steroids or CYP450 enzyme-inducing anticonvulsants.
* Subjects must have a LVEF ≥ 50% or ≥ lower limit of normal for the institution based on MUGA scan or ECHO. The same method of cardiac evaluation must be used consistently throughout the study.
* Subjects in the expanded cohort phase must have archived tumor tissue samples available for biomarker analysis. It is preferable that a paraffin-embedded tissue block from archived tumor tissue from the primary tumor be submitted.
* Subjects must provide informed consent and blood samples to the pharmacogenetics research.
* Subjects must be able to swallow and retain oral medications.
* Subjects must have adequate hematological, hepatic, and renal function as defined: Hematologic: absolute neutrophil count (ANC) ≥1.5 X 10^9/L, hemoglobin ≥10 g/dL, platelets ≥100 X 10^9/L; Hepatic: serum bilirubin≤ upper limit of normal (ULN), AST and ALT ≤ 5 x ULN if documented liver metastases, AST and ALT ≤ 3 X ULN without liver metastases; Renal: calculated creatinine clearance ≥50 mL/min.
* A female is eligible to enter and participate in this study if she is of:
* Non-childbearing potential (i.e., women with functioning ovaries who have a current documented hysterectomy, or bilateral tubal ligation, or women who are post-menopausal defined as documented absence of menses for > 12 months or women with a documented bilateral oophorectomy);
* Childbearing potential (i.e. women with functioning ovaries and no documented impairment of oviductal or uterine function that would cause sterility.) This category includes women with oligomenorrhoea (severe), women who are perimenopausal, and young women who have begun to menstruate. These subjects must have a negative serum pregnancy test at Screening (≤7 days prior to administration of first dose of investigational product), and agree to use adequate contraception beginning at least 2 weeks prior to the first does of investigational product and for 28 days after the final dose of investigational product. GSK acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows:
* An intrauterine device with a documented failure rate of less than 1% per year.
* Vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.
* Complete abstinence from sexual intercourse for 14 days before exposure to investigation product, through the clinical trial, and for at least 28 days after the last dose of investigational product.
* Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide).
* Oral contraceptives are not reliable due to potential drug-drug interaction.
* Male subjects with a female partner of childbearing potential are eligible to enter and participate in the study if they practice adequate barrier methods of contraception (see above) or abstinence during the study from the first dose of investigational product until 3 months after the final dose of investigational product.

Exclusion Criteria:

* Subjects who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to the first dose of investigational product or who have unresolved or unstable, serious toxicity from prior administration of another investigational drug and/or of prior cancer treatment.
* Subjects who have received an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of investigational product.
* Subjects taking prohibited medications listed in the protocol.
* Subjects with a known immediate or delayed hypersensitivity or untoward reaction to topotecan or other related compounds, or to drugs chemically related to lapatinib. These include other anilinoquinazolines, such as gefitinib, erlotinib, or other chemically-related compounds.
* Subjects with presence of uncontrolled infection.
* Subjects with malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel.
* Subjects with uncontrolled or symptomatic angina, arrhythmias.
* Subjects with Class II to IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Women who are pregnant or lactating.
* Subjects who have received an allogeneic bone marrow transplant.
* Subjects with any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study.
* Subjects with psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Subjects with clinical history, current alcohol or illicit drug use which, in the judgment of the investigator, would interfere with the subject's ability to comply with the dosing schedule and protocol-specified evaluations.
* Subjects with current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
The maximum-tolerated dose (MTD) regimen of the combination will be defined as the maximum dose level at which no more than one subject out of six experiences a dose-limiting toxicity (DLT) after completing one treatment cycle. | Study cancelled prior to FCI.

SECONDARY OUTCOMES:
Adverse events and changes from baseline in laboratory values, ECGs, Multiple gated Acquisition (MUGA) scanning/Echocardiogram (ECHO), and vital signs will be evaluated to assess safety and tolerability. | Study cancelled prior to FCI.
Topotecan pharmacokinetic parameters may include AUC(0-∞), AUC(0-τ), Cmax, tmax, t½, and tlag, | Study cancelled prior to FCI.
alone and in combination with lapatinib. Lapatinib pharmacokinetic parameters may include AUC(0-τ), Cτ, Cmax, tmax, and tlag, alone and in combination with topotecan. | Study cancelled prior to FCI.
Disease assessments will be obtained every two cycles and will be recorded as tumor response (e.g. complete response [CR], partial response [PR], stable disease [SD], or progressive disease [PD]). | Study cancelled prior to FCI.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Philadelphia, Pennsylvania